CLINICAL TRIAL: NCT00705133
Title: Using Either Intravenous (IV) or Subcutaneous (SQ) Treprostinil to Treat Pulmonary Hypertension Related to Underlying Interstitial Lung Disease
Brief Title: Treprostinil Therapy For Patients With Interstitial Lung Disease And Severe Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rajan Saggar (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Rajan Saggar, Principal Investigator, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-11-087-01
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Pulmonary Arterial Hypertension; Interstitial Lung Disease; Idiopathic Pulmonary Fibrosis
Keywords: pulmonary hypertension; pulmonary fibrosis; interstitial lung disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis; Hypertension, Pulmonary; Pulmonary Fibrosis | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treprostinil-treated (Experimental): Patients with pulmonary fibrosis with an advanced pulmonary hypertension phenotype will be treated with parenteral treprostinil in an open-label fashion
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — For both SQ and IV routes, treprostinil will be started in the hospital at 1ng/kg/min and titrated up by 1ng/kg/min every 1-3 days as tolerated
  Other Names: remodulin

SUMMARY:
Our hypothesis is that IV or SQ Treprostinil can improve 6 minute walk distance, hemodynamics and quality of life in patients with interstitial lung disease and severe secondary pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Patients with pulmonary hypertension (PH) complicating pulmonary fibrosis are at increased risk of death. There are no therapies proven to be effective in this population, targeting the pulmonary hypertension. The purpose of this study is to evaluate parenteral treprostinil in an open-label fashion in patients with pulmonary fibrosis and an advanced PH phenotype.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must have IPF and severe pulmonary arterial hypertension (PAH) documented on standard of care right-heart catheterization (RHC) and planned to receive therapy with treprostinil as recommended by the treating physician.

1. All subjects must have high resolution CT scan (HRCT) diagnostic of IPF (performed as part of standard of care evaluation) or if available, biopsy proven histological usual interstitial pneumonia (UIP).
2. Severe pulmonary arterial hypertension defined as a resting mean pulmonary artery pressure (mPAP) > 35 mm Hg; AND pulmonary vascular resistance (PVR) > 3 woods-units; AND pulmonary capillary wedge pressure (PCWP) < 18 mm Hg by right-heart catheterization (RHC) performed as part of standard of care evaluation.
3. All subjects must be planned to receive treprostinil therapy as recommended by their treating physician.

Exclusion Criteria:

1. Acute or chronic impairment other than dyspnea (e.g. angina pectoris, intermittent claudication) limiting the ability to perform standard of care six-minute walk tests (6MWT).
2. Six-minute walk distance (6MWD) < 50 meters at screening or baseline standard of care evaluations
3. Standard of care pulmonary function test (PFT) showing forced expiratory volume in one second (FEV1)/ forced vital capacity (FVC) ratio < 0.65
4. Standard of care pulmonary function test (PFT) showing a residual volume >120% predicted
5. Standard of care high-resolution chest computed tomography (HRCT) showing emphysema extent > 30%
6. Any investigational therapy as part of a clinical trial for any indication with 30 days before screening
7. Change in dose of treatment for IPF - investigational agent (gamma interferon-1b, pirfenidone, etanercept, and any other investigational agent intended to treat IPF), corticosteroids, or cytotoxic agents, within 30 days before screening. That is, subjects can be on any of these agents provided the dose is stable for at least 30 days prior to enrollment.
8. Current treatment for pulmonary hypertension with other prostaglandins (epoprostenol or iloprost)
9. Change in dose of treatment for PAH - (bosentan, sitaxsentan, ambrisentan, tadalafil, sildenafil, vardenafil, calcium channel blockers, nitrates, digitalis), within 30 days before screening. That is, subjects can be on any of these agents provided the dose is stable for at least 30 days prior to enrollment
10. Pulmonary rehabilitation initiated within 30 days of baseline.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, MD, Principal Investigator — David Geffen School of Medicine, UCLA; David Zisman, MD, Principal Investigator — David Geffen School of Medicine, UCLA
Locations (1):
- David Geffen School of Medicine, UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saggar R, Khanna D, Vaidya A, Derhovanessian A, Maranian P, Duffy E, Belperio JA, Weigt SS, Dua S, Shapiro SS, Goldin JG, Abtin F, Lynch JP 3rd, Ross DJ, Forfia PR, Saggar R. Changes in right heart haemodynamics and echocardiographic function in an advanced phenotype of pulmonary hypertension and right heart dysfunction associated with pulmonary fibrosis. Thorax. 2014 Feb;69(2):123-9. doi: 10.1136/thoraxjnl-2013-204150. PMID 24431095

RESULTS

PARTICIPANT FLOW:
Groups:
- Treprostinil-treated: Patients with pulmonary fibrosis with an advanced pulmonary hypertension phenotype will be treated with parenteral treprostinil in an open-label fashion
  Treprostinil: For both subcutaneous (SQ) and IV routes, treprostinil will be started in the hospital at 1ng/kg/min and titrated up by 1ng/kg/min every 1-3 days as tolerated
Period: Overall Study
Arm/Group | Treprostinil-treated
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treprostinil-treated
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: 6 Minute Walk Distance
Description: American Thoracic Society (ATS) Practice Guideline based 6-minute walk (6MW) distance
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treprostinil-treated
Number analyzed (Participants) | 15
meters | 230 (114)

2. Secondary Outcome: Pulmonary Vascular Resistance
Description: repeat right heart catheterization
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: wood units
Arm/Group | Treprostinil-treated
Number analyzed (Participants) | 15
wood units | 496 (229)

3. Secondary Outcome: SF-36 Quality of Life
Description: SF-36 physical component summary (PCS) which is one component of the SF-36 survey. The health assessment questionnaire Short Form 36 Version 2.0 (SF-36 V2 ) determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary score (PCS) of the SF-36. Scores on each item are summed and averaged (range = 0 "worst"-100 "best").
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treprostinil-treated
Number analyzed (Participants) | 15
score on a scale | 28 (8.8)

4. Secondary Outcome: Brain Natriuretic Peptide
Description: brain natriuretic peptide (BNP) is a measure of right ventricular distension and/or stress due to pressure or volume overload
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treprostinil-treated
Number analyzed (Participants) | 15
pg/mL | 228 (340)

ADVERSE EVENTS:
Arm/Group | Treprostinil-treated
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil-treated (N=15)
general prostacyclin adverse reaction profile (Gastrointestinal disorders) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No